CLINICAL TRIAL: NCT00860366
Title: Randomized, Double Blind Study Assessing the Clinical Efficacy of Combined Treatment With Uric Acid and rtPA Administered Intravenously in Acute Ischemic Stroke Patients Within the First 4.5 Hours of Symptoms Onset
Brief Title: Efficacy Study of Combined Treatment With Uric Acid and rtPA in Acute Ischemic Stroke
Acronym: Urico-Ictus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Angel Chamorro, MD (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Angel Chamorro, MD, MD, PhD, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URICOICTUS-1-2007; EudraCT 2007-002687-95; FIS EC07-90276
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; thrombolysis; alteplase; uric acid; neuroprotection; oxidative stress
MeSH Terms: conditions — Ischemic Stroke | interventions — Uric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uric Acid (Experimental): Single intravenous infusion of 1 gram of Uric Acid dissolved in vehicle (500 ml of 0'1% Lithium Carbonate and 5% Mannitol).
  Interventions: Drug: Uric Acid
- Vehicle (Placebo Comparator): Single intravenous infusion of a 500 ml vehicle containing 0'1% Lithium Carbonate and 5% Mannitol.
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Uric Acid — 1 gram dissolved in a vehicle containing 500 ml of 0'1% Lithium Carbonate and 5% Mannitol, IV (in the vein), single dose.
  Arms: Uric Acid
Other: Vehicle — Single intravenous infusion of a 500 ml vehicle containing 0'1% Lithium Carbonate and 5% Mannitol.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether the combined treatment with Uric Acid and rtPA is superior to rtPA alone in terms of clinical efficacy in acute ischemic stroke patients treated within the first 4.5 hours of symptoms onset.

DETAILED DESCRIPTION:
Oxidative stress is a major contributor to brain damage in patients with ischemic stroke. Uric acid (UA) is an endogenous product derived from the metabolism of purins which in man is responsable of the 60% of the total antioxidant capacity of the organism. Recent experimental evidences gathered by our and other research groups have shown that the exogenous administration of UA is neuroprotective both in cortical and subcortical brain areas as the result of its antioxidant properties. In these studies, animals treated with UA disclosed smaller brain infarction after transient focal ischemia, both using the intraluminal model or after the injection of autologous clots. Moreover, our group first described greater neuroprotection in animals pretreated with rtPA (alteplase). Likewise, we have recently shown that the administration of UA was free of serious adverse effects in stroke patients receiving rtPA within 3 hours of stroke onset. Yet, preliminary data suggested that this intervention might translate into clinical benefits at 3 months follow-up. Based on these data, we aim to conduct a phase 3, randomized, double-blind, controlled trial assessing the clinical efficacy of UA administration in acute ischemic stroke patients. Currently, rtPA is the only approved therapy for stroke patients within the first hours of clinical onset, and oxidative stress is thought particularly relevant following ischemia/reperfusion. Based on this ground, we aim to conduct this phase 3 clinical trial in ischemic stroke patients which are currently treated with rtPA within the 4'5 hour window.

ELIGIBILITY:
Inclusion criteria:

* Age older than 18 years old.
* Acute ischemic stroke treated with rtPA within the first 4.5 hours of clinical onset. Baseline National Institute of Health Stroke Scale (NIHSS) >6 and <25, and modified Rankin Scale (mRS) of 2 prior to the stroke.
* Cranial CT disclosing the absence of blood in the CNS.
* Informed consent.

Exclusion criteria:

* Presence of any of the valid exclusion criteria for the administration of rtPA in the current clinical practise.
* History of gout with or without history of gouty nephropathy, or uric lithiasis. Asymptomatic hiperuricemia under chronic treatment with allopurinol, or chronic treatment with lithium.
* Chronic renal insufficiency (baseline creatinine > 1,5mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a mRS of 0 to 1 at 3 months after treatment, or 2 in those patients with a mRS 2 prior to the inclusion in the study | 90 days after the inclusion.

SECONDARY OUTCOMES:
Proportion of patients with NIHSS <2 at 2 hours after completing the experimental treatment. | 2 hours after completing the experimental treatment
Proportion of patients with NIHSS <1 at day 90. | Day 90
Proportion of patients achieving a Barthel scale of 95 to 100 at day 90 | Day 90
All-cause mortality within the first 90 days. | Day 90
Final Infarction Volume measured by means of MRI or multimodal CT at 72 hours of onset (in specific centers) | 72 hours
Proportion of patients with an intracranial hemorrhage associated to a worsening of 4 points in the NIHSS within the first 36 hours of treatment. | 36 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Chamorro, MD, PhD., Study Director — Comprehensive Stroke Center, Hospital Clínic Barcelona, Spain.
Locations (10):
- Spain (10):
  - Hospital General Universitario de Albacete, Albacete, Albacete
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu y Sant Pau, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Bellvitge, Barcelona
  - Corporació Sanitària del Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Dr Josep Trueta, Girona, Girona
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid

REFERENCES:
- [Background] Chamorro A, Obach V, Cervera A, Revilla M, Deulofeu R, Aponte JH. Prognostic significance of uric acid serum concentration in patients with acute ischemic stroke. Stroke. 2002 Apr;33(4):1048-52. doi: 10.1161/hs0402.105927. PMID 11935059
- [Background] Chamorro A, Planas AM. Yin and yang of uric acid in patients with stroke. Stroke. 2004 Jan;35(1):e11-2; author reply e11-2. doi: 10.1161/01.STR.0000107762.79571.7D. Epub 2003 Dec 11. No abstract available. PMID 14671231
- [Background] Chamorro A, Planas AM, Muner DS, Deulofeu R. Uric acid administration for neuroprotection in patients with acute brain ischemia. Med Hypotheses. 2004;62(2):173-6. doi: 10.1016/S0306-9877(03)00324-4. PMID 14962621
- [Background] Romanos E, Planas AM, Amaro S, Chamorro A. Uric acid reduces brain damage and improves the benefits of rt-PA in a rat model of thromboembolic stroke. J Cereb Blood Flow Metab. 2007 Jan;27(1):14-20. doi: 10.1038/sj.jcbfm.9600312. Epub 2006 Apr 5. PMID 16596120
- [Background] Amaro S, Soy D, Obach V, Cervera A, Planas AM, Chamorro A. A pilot study of dual treatment with recombinant tissue plasminogen activator and uric acid in acute ischemic stroke. Stroke. 2007 Jul;38(7):2173-5. doi: 10.1161/STROKEAHA.106.480699. Epub 2007 May 24. PMID 17525395
- [Background] Amaro S, Planas AM, Chamorro A. Uric acid administration in patients with acute stroke: a novel approach to neuroprotection. Expert Rev Neurother. 2008 Feb;8(2):259-70. doi: 10.1586/14737175.8.2.259. PMID 18271711
- [Background] Amaro S, Chamorro A. Translational stroke research of the combination of thrombolysis and antioxidant therapy. Stroke. 2011 May;42(5):1495-9. doi: 10.1161/STROKEAHA.111.615039. Epub 2011 Apr 7. PMID 21474803
- [Background] Amaro S, Urra X, Gomez-Choco M, Obach V, Cervera A, Vargas M, Torres F, Rios J, Planas AM, Chamorro A. Uric acid levels are relevant in patients with stroke treated with thrombolysis. Stroke. 2011 Jan;42(1 Suppl):S28-32. doi: 10.1161/STROKEAHA.110.596528. Epub 2010 Dec 16. PMID 21164140
- [Derived] Amaro S, Renu A, Laredo C, Castellanos M, Arenillas JF, Llull L, Rudilloso S, Urra X, Obach V, Chamorro A; on behalf of the URICO-ICTUS investigators. Relevance of Collaterals for the Success of Neuroprotective Therapies in Acute Ischemic Stroke: Insights from the Randomized URICO-ICTUS Trial. Cerebrovasc Dis. 2019;47(3-4):171-177. doi: 10.1159/000500712. Epub 2019 Jun 4. PMID 31163434
- [Derived] Chamorro A, Amaro S, Castellanos M, Gomis M, Urra X, Blasco J, Arenillas JF, Roman LS, Munoz R, Macho J, Canovas D, Marti-Fabregas J, Leira EC, Planas AM; URICO-ICTUS Investigators. Uric acid therapy improves the outcomes of stroke patients treated with intravenous tissue plasminogen activator and mechanical thrombectomy. Int J Stroke. 2017 Jun;12(4):377-382. doi: 10.1177/1747493016684354. Epub 2016 Dec 20. PMID 28345429
- [Derived] Amaro S, Laredo C, Renu A, Llull L, Rudilosso S, Obach V, Urra X, Planas AM, Chamorro A; URICO-ICTUS Investigators. Uric Acid Therapy Prevents Early Ischemic Stroke Progression: A Tertiary Analysis of the URICO-ICTUS Trial (Efficacy Study of Combined Treatment With Uric Acid and r-tPA in Acute Ischemic Stroke). Stroke. 2016 Nov;47(11):2874-2876. doi: 10.1161/STROKEAHA.116.014672. Epub 2016 Oct 6. PMID 27758945
- [Derived] Llull L, Laredo C, Renu A, Perez B, Vila E, Obach V, Urra X, Planas A, Amaro S, Chamorro A. Uric Acid Therapy Improves Clinical Outcome in Women With Acute Ischemic Stroke. Stroke. 2015 Aug;46(8):2162-7. doi: 10.1161/STROKEAHA.115.009960. Epub 2015 Jul 9. PMID 26159792
- [Derived] Chamorro A, Amaro S, Castellanos M, Segura T, Arenillas J, Marti-Fabregas J, Gallego J, Krupinski J, Gomis M, Canovas D, Carne X, Deulofeu R, Roman LS, Oleaga L, Torres F, Planas AM; URICO-ICTUS Investigators. Safety and efficacy of uric acid in patients with acute stroke (URICO-ICTUS): a randomised, double-blind phase 2b/3 trial. Lancet Neurol. 2014 May;13(5):453-60. doi: 10.1016/S1474-4422(14)70054-7. Epub 2014 Apr 2. PMID 24703208